CLINICAL TRIAL: NCT00356772
Title: Comparison of Azithromycin Level in Tears and in Conjunctiva After Repeated Instillations of T1225 1.5% Eye Drops or After a Single Per Os Administration of Zithromax® (Azithromycin 1g), in 36 Healthy Volunteers
Brief Title: Azithromycin Level in Tears and in Conjunctiva in 36 Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Laboratoires Thea (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LT1225-PI4-11/02(F)
Record Dates: First submitted 2006-07-25; First posted 2006-07-26 (Estimated); Last update posted 2006-07-26 (Estimated); Status verified 2006-07

CONDITIONS: Eye Infections, Bacterial
MeSH Terms: conditions — Eye Infections, Bacterial | interventions — Azithromycin

INTERVENTIONS:
Drug: Azithromycin

SUMMARY:
To evaluate azithromycin ocular conjunctiva concentrations 7 and 14 days after treatment initiation.

To assess ocular and systemic tolerance/safety and azithromycin tear concentrations on Day 7

DETAILED DESCRIPTION:
The aim of the present study was to compare azithromycin tear and conjunctival ocular concentrations after one instillation of T1225 1.5% eye drops, twice a day during one day versus one instillation of T1225 1.5% eye drops, twice a day during 3 days versus an oral single dose of 1g azithromycin.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent;
* Healthy volunteers;
* Registered in the national register of healthy volunteers;
* Male or female aged from 18 to 45 years old;
* Able to understand the study instructions;
* Likely to comply with the study schedule and treatment;
* Normal subjective ocular symptoms, Schirmer test > 10 mm in 5 min and corrected visual acuity >= 6/10 in both eyes

Exclusion Criteria:

* Ocular trauma, infection or inflammation within the last 3 months;
* Blepharitis;
* Conjunctival hyperaemia (score >= 2);
* Fluorescein-stained punctuations (score >= 1b);
* Hypersensitivity to one of the products used in the study;
* Clinically relevant allergy;
* Medical or surgical history incompatible with the study;
* Recent acute illness;
* Ocular surgery, including LASIK, LASEK and PRK within the last 12 months;
* Other ocular lasers or Zithromax® or Azadose® within the last 3 months;
* Systemic antibiotics and ocular medications within the last month;
* Contact lenses within the last week;
* Any medication on Day 0 and during the study (except paracetamol and contraceptives).

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Dates: Start 2003-02; Study Completion 2003-03

PRIMARY OUTCOMES:
Azithromycin Ocular Conjunctiva Concentrations on Days 7 and 14.
Azithromycin Tear Concentrations on Day 7.

SECONDARY OUTCOMES:
Tolerance

CONTACTS AND LOCATIONS:
Overall Officials: Claude DUBRAY, Professor, Principal Investigator — Centre de Pharmacologie Clinique - Clermont-Ferrand (France)